CLINICAL TRIAL: NCT05757752
Title: Mind Body Program for Vascular Disease Proof-of-Concept Study
Brief Title: Mind Body Program for Vascular Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000034225
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Participants meeting eligibility criteria will participate in the Mind Body Program for Vascular Disease, working in-person or via telehealth with a study interventionist for an hour weekly in 6-8 week cycles learning problem-solving techniques targeting mood/distress and enhancing disease management strategies. Participants will be assessed at baseline, 3-months, and 6-months.
  Interventions: Behavioral: Problem Solving Therapy and Integrated Care

INTERVENTIONS:
Behavioral: Problem Solving Therapy and Integrated Care — The intervention, will consist of problem solving therapy techniques to promote PAD self-management behaviors and depression/distress management.

SUMMARY:
The purpose of the current study is to conduct a proof-of-concept test regarding the delivery of a Mind Body Program for vascular disease, focusing on support for depression, stress, and adherence, as part of patients' chronic disease management for peripheral artery disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Rutherford score 1-4 (mild-severe claudication, or ischemic rest pain)
* Resting ankle-brachial index assessment ≤0.90 or drop in post-exercise ankle pressure ≥20 mmHg or non-compressible ankle-brachial index (≥1.30) or toe brachial index less than 0.70 in the past year
* Positive depression screening result (positive PHQ-9 result ≥10) or high stress screening result (10-item Perceived Stress Scale Score ≥27)

Exclusion Criteria:

* Not speaking either English or Spanish
* Age ≥18 years
* Currently incarcerated
* Current alcohol dependency or other substance use disorder (score ≥ 5 on NM-ASSIST)
* Cognitive impairment (T-MoCA Short <10)
* Acute suicidal risk (positive screen ASQ Tool)
* History of psychosis or bipolar disorder
* Previously enrolled in the study
* Unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in PAD-Specific Health Status on the Peripheral Artery Questionnaire (PAQ) | Baseline and 6months.
  The PAQ Summary Score is a 20-item, validated, self-report instrument quantifying patients' disease specific health status. The measure is comprised of 6 domains including physical limitations, symptoms, symptom stability, social functioning, treatment satisfaction, and quality of life. Total scores range from 0 to 100, with higher scores indicate better functioning. Change will be determined using comparisons between baseline and 6 months.
Change in Depressive Symptoms assessed by Symptom Checklist-20 (SCL-20) | Baseline, 3months, and 6months.
  Patient depressive symptoms will be measured using the SCL-20. The SCL-20 is a 20-item, validated, self-report instrument assessing depressive symptom intensity. Total scores range from 0 to 80, with higher score indicating higher depressive symptom intensity. Change will be determined using comparisons between baseline, 3 months and 6 months.
Change in Depressive Symptoms assessed by Patient Health Questionnaire (PHQ-9) | initial screening, baseline, 3months, and 6months
  Patient depressive symptoms will be measured using the 9-item PHQ-9. PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-45. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety. Change will be determined by whether sufficient improvement is demonstrated between initial screening, baseline, 3 months, and 6 months. Sufficient improvement is defined as a 30% improvement if the prior depression score was between 5-10, or a 50% improvement if the score was greater than 20.
Change in Stress Symptoms assessed using Perceived Stress Scale (PSS-10) | initial screening, baseline, 3months, and 6months.
  Patient distress levels will be measured using the 10-item PSS-10. The PSS-10 is a 10-item, validated, self-report, questionnaire used to assess perceived control and confidence in managing stressful situations over the past month. Scores range from 0 to 40, with higher scores indicated higher levels of perceived stress. Change will be determined by whether sufficient improvement is demonstrated between initial screening up to 6 months. Sufficient improvement is defined as moving from a high stress (score 27-40 on PSS-10) to a moderate stress (score 14-26).

SECONDARY OUTCOMES:
Change in Care Satisfaction using COPES Satisfaction with Depression Question | baseline and 6months
  Patient satisfaction with the care they receive participating in the Mind Body Program for Vascular Disease will be measures using the single item COPES Satisfaction with Depression Question. This item asks patients to rate the quality of professional care they have received for their symptoms of distress or depression over the last 2 months. Scores range from 1 (Excellent) to 5 (Poor), with higher scores indicating worse satisfaction. Patients who did not receive care for distress or depression symptoms have the option to indicate this as their response. Change will be determined using comparisons between baseline and 6 months.

OTHER OUTCOMES:
Change in Physical activity using step count | baseline, 3months, and 6months
  Physical activity levels will be measured as 7-day averaging of step counts by Garmin Vivofit activity trackers. Sedentary behavior is defined as <7000 steps per day and being physically active is defined as ≥7000 steps per day. The investigators will consider a clinically meaningful treatment signal that >50% of patients will display active behavior (7-day average of ≥7000 steps/day) at 6 months.
Change in Physical activity using Walking Impairment Questionnaire | baseline, 3months, and 6months
  The Walking Impairment Questionnaire is a 19-item, validated, self-report measure of the degree of difficulty participants experience related to walking distance and speed, as well as symptoms they experience while walking (e.g., stiffness, pain, aches). Scores range from 0-100 with lower scores indicating lower performance. Change will be determined using comparisons between baseline up to 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Health Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No